CLINICAL TRIAL: NCT03633513
Title: Inflammatory Parkinson's Disease (PD) Clinical Biomarker Profiling in T Cells
Brief Title: Parkinson's Disease Inflammatory Biomarker Profiling
Status: Terminated | Type: Observational
Why Stopped: COVID-19
Sponsor: Longevity Biotech (Industry)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); Corporal Michael J. Crescenz VA Medical Center - Philadelphia (Unknown)
Responsible Party: Sponsor
Other Study IDs: LBT-PD-003
Record Dates: First submitted 2018-07-15; First posted 2018-08-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Parkinson Disease
Keywords: Immune System; Immunology; Neuroinflammation; Inflammation; Neuroprotection
MeSH Terms: conditions — Parkinson Disease; Neuroinflammatory Diseases; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: US Export: No

GROUPS / COHORTS (2):
- Patients: Clinical diagnosed Parkinson's disease patients
  Interventions: Diagnostic Test: LBT-3627; Diagnostic Test: Immunological profiling
- Caregivers: Environmentally matched healthy control subjects
  Interventions: Diagnostic Test: LBT-3627; Diagnostic Test: Immunological profiling

INTERVENTIONS:
Diagnostic Test: LBT-3627 — Immunomodulatory agent
Diagnostic Test: Immunological profiling — Comprehensive profiling of inflammatory and anti-inflammatory markers (incl. cellular, molecular) including cellular functional assays

SUMMARY:
This study compares a comprehensive panel of immunological biomarkers between Parkinson's disease patients and healthy, environmentally matched participants. This unique study design provides the ability to control for differences in environment between study subjects. The goal of this study is to 1) identify a specific set of immunological markers that correlate with a clinical diagnosis of Parkinson's disease and 2) stratify patients by disease severity using these same biomarkers.

ELIGIBILITY:
Inclusion Criteria

All Participants

* Subjects must be willing and able to participate in study
* Subjects must be willing and able to provide written consent to participate.
* Subjects must be willing and able to comply with scheduled clinic visits and study procedures (UPDRS exam, blood draw and complete a questionnaire)
* Subjects are not currently taking an immunomodulatory (e.g. anti- tumor necrosis factor (TNF), immunosuppressants/stimulants) agent in the past 90 days
* No active or recent (< 3 weeks) infection requiring clinical intervention and/or pharmaceutical treatment or febrile neutropenia within the last week.
* 18-89 years old

Parkinson's Disease Patients

* Clinical diagnosis of PD by a movement disorders specialist consistent with standard criteria
* Able to attend a clinical visit in the 'off' state
* Hoehn and Yahr stage I-IV

Caregiver Controls

• Individuals without PD who share environmental exposures (i.e. spouses, children, caregivers or other individuals who frequently spend significant time (>6 hours) in proximity to the PD subject) OR age and sex matched healthy individuals from general population

Exclusion Criteria

All Participants

* Unstable cardiopulmonary or cerebrovascular disease
* Renal disease or failure w/ serum creatinine greater than 2.5
* Severe or unstable depression or other axis I psychopathology
* Epilepsy
* Prior brain surgery related to PD (DBS, cell implantation, gene therapy, etc.)
* Severe head injury with evidence of brain injury
* Essential Thrombocythemia (ET) (>450,000 platelets/mL)
* Patients currently being treated with any of the following, within the past 5 days:
* Immunomodulatory agents (e.g. Remicade®, Humira®, Enbrel®) (within the past 90 days)
* Corticosteroids
* Probenecid®
* Coenzyme Q10®
* Anticoagulants

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with Parkinson's disease and their caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-03-13 (Actual); Study Completion 2020-03-13 (Actual)

PRIMARY OUTCOMES:
Unified Parkinson Disease Rating Scale | 1 hour
  Clinical scoring system to evaluate severity of Parkinson's disease in patients

SECONDARY OUTCOMES:
Interleukin-17 | 48 hours
  Proinflammatory cytokine
FoxP3 | 48 hours
  Regulatory Tcell marker
GM-CSF | 48 hours
  Cytokine
LRRK2 | 48 hours
  Leucine rich region kinase 2 protein
VPAC2 | 48 hours
  Regulates TH1/TH2 balance of inflammatory system
Interferon gamma | 48 hours
  Inflammatory cytokine
Tumor necrosis factor alpha | 48 hours
  Inflammatory cytokine

OTHER OUTCOMES:
Immune cell functional analysis | 1 week
  Performance evaluation of protective immune cells (Tregs) compared to responder immune cells (Tresp)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Shandler, PhD, Principal Investigator — Longevity Biotech, Inc
Locations (2):
- United States (2):
  - Corporal Michael J. Crescenz VA Medical Center, Philadelphia, Pennsylvania
  - Longevity Biotech, Inc, Philadelphia, Pennsylvania

REFERENCES:
- See also: Michael J. Fox Trial Finder — https://foxtrialfinder.michaeljfox.org/trial/5308/